CLINICAL TRIAL: NCT02919722
Title: The Effects of Playing Live Music in Music Therapy/Occupational Therapy Co-treatment on Unilateral Spatial Neglect
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-00189
Record Dates: First submitted 2016-09-28; First posted 2016-09-29 (Estimated); Last update posted 2020-08-19 (Actual); Status verified 2020-08

CONDITIONS: Unilateral Spatial Neglect (USN)
Keywords: Music therapy; sensorimotor cortex; brain injury
MeSH Terms: conditions — Brain Injuries | interventions — Music Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Music interventions (Experimental): Live music will be provided on the patient's neglected side and patients will be encouraged to play music interactively with a focus towards that side whenever possible
  Interventions: Behavioral: Music Therapy

INTERVENTIONS:
Behavioral: Music Therapy — The majority of each study session will be spent engaging in music therapy: playing live music with a music therapist with the help of an occupational therapist. At the beginning and end of each session subjects will complete 2 assessments.

SUMMARY:
Investigators hypothesize, based on anecdotal evidence to date, that active music making interventions conducted on a patient's neglected side will result in improved attention to that side and that this will be measurable within session.

DETAILED DESCRIPTION:
An open, single group of ten patients selected will receive a 30 minute music therapy/occupational therapy co-treatment intervention. Music interventions will be performed by a licensed, Board-Certified Music Therapist while a licensed Occupational Therapist will provide support, assistance, and measurements of behavioral attention/inattention. At the outset of the first session patients will be briefly, informally interviewed to ascertain their musical preferences, which will then be integrated into the music therapist's interventions whenever possible to maximize engagement and therapeutic rapport. Live music will be provided on the patient's neglected side and patients will be encouraged to play music interactively with a focus towards that side whenever possible. An outcome measurement tool (Star Cancellation Test) will be focused on measuring hemispheric neglect and administered at the beginning and end of each session to measure within session changes.

ELIGIBILITY:
Inclusion Criteria:

* Patients experiencing unilateral left spatial neglect post brain injury (stroke, TBI, N-TBI).
* Patients able to follow two step commands and maintain attention to task for five minutes in a quiet environment.
* The KF-NAP, which is administered to all patients with suspected neglect on admission, will be used as a screening tool for the neglect syndrome. Inclusion criteria will be participants with score of ≤ 5.
* Patients must be able to hold a pencil to complete the SCT
* Patients must be able to discriminate between distractor items (words versus big and small stars) and see items in picture cards
* Patients communicate willingness to participate in music therapy interventions.
* Admission to acute inpatient rehabilitation unit at NYU/HJD.
* Patient will have the ability to provide informed consent.

Exclusion Criteria:

* Visual impairment.
* Right side or dominant hand impairment.
* Any social or medical problem that precludes completion of the protocol.
* Patients who have sensory neglect or motor neglect , as the SCT cannot be used with this population
* Severe language comprehension impairment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2019-12-19 (Actual); Study Completion 2019-12-19 (Actual)

PRIMARY OUTCOMES:
Star Cancellation Test and Picture Scanning Test (from the Behavioral Inattention Test (BIT) | 1 Day
  54 targets dispersed amongst 75 distractors. Patients are asked to cross out all of the small stars within the field, placed at midline, using a pen.
Picture Scanning Test (PST) | 1 Day
  3 large color photos that depict: (1) a meal on a dish, (2) a wash basin and toiletries, (3) a large window flanked by sundry objects. Participant is asked to name and point to the main items see in the picture.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Im, MD, Principal Investigator — New York University Medical School
Locations (1):
- New York University School of Medicine, New York, New York, United States